CLINICAL TRIAL: NCT03328624
Title: A Preliminary Clinical Usability Study to Assess Design, Comfort, Wearability, and Acceptance of Recovery Force's Deep Vein Thrombosis (DVT) Cuff
Brief Title: A Preliminary Clinical Usability Study for the Recovery Force DVT II Cuff
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Recovery Force LLC (Industry)
Responsible Party: Principal Investigator, David Armstrong, Professor of Surgery and Director, Southwestern Academic Limb Salvage Alliance (SALSA), University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS-17-00865
Record Dates: First submitted 2017-10-09; First posted 2017-11-01 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Deep Vein Thrombosis; Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- DVT Cuff users (Experimental): Current or previous DVT cuff users
  Interventions: Device: Deep Vein Thrombosis (DVT) Cuff

INTERVENTIONS:
Device: Deep Vein Thrombosis (DVT) Cuff — Recovery Force's DVT II Cuff
  Other Names: RF1400

SUMMARY:
A preliminary clinical usability study to assess design, comfort, wearability, and acceptance of Recovery Force's Deep vein thrombosis (DVT) cuff

DETAILED DESCRIPTION:
A single site, observational study will be conducted at the University of Southern California (USC) with participants who have and/or have had previous experience with DVT pneumatic cuffs. Study staff will examine participants overall experience, product functionality and perceived adherence to Recovery Force's DVT II cuff.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Age 18-65 who have had exposure with a DVT cuff on the calf within the last 6 months from a previous or current clinical condition

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, MD, PhD, Principal Investigator — Professor of Surgery and Director, SALSA@USC
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DVT Cuff Users
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DVT Cuff Users
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 22
  More than one race | 8
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Comfort and Patient Acceptance
Description: 1. FULL SCALE NAME: Wearability, comfort, and acceptance of the DVT cuff Scale. Created a likert-type scale in RedCAP with values from 0 to 10, with higher score equaling better outcome.
  2. TIME FRAME: Each participant wore the DVT cuff under study for 20 minutes, and evaluated their experience using the scale above.
  Evaluated through User Questionnaire: Recovery Force DVT Cuff - Post-Demonstration Patient Questionnaire; and subject interview
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DVT Cuff Users
Number analyzed (Participants) | 36
score on a scale | 8.89 (1.77)

ADVERSE EVENTS:
Time Frame: 1 day
Description: Single-use study of DVT cuff
Arm/Group | DVT Cuff Users
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT03328624/Prot_SAP_000.pdf